CLINICAL TRIAL: NCT05689112
Title: Microscopy Imaging of Whole-mount Stained Human Tissues: Development of an Imaging Platform for Intraoperative Tumor Margin Delineation
Brief Title: Microscopy Imaging of Whole-mount Stained Human Tissues
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211038RINA
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-01

CONDITIONS: Tumor, Brain; Tumor, Breast; Tumor Skin
Keywords: intraoperative assessment; whole-mount H&E staining; surgical border assessment
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this clinical trial is to develop an imaging platform for intraoperative tumor margin delineation in 250 cases of tumor-suffered patients. The main questions it aims to answer are:

• to develop the protocol of rapid assessment of surgical specimens without need for fixation, embedding, and cryosectioning required for conventional histopathology.

Participants will provide a small piece of their surgical specimens from tumor removal surgery .

If there is a comparison group: Researchers will compare normal specimens to see if we can observe the difference.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are more than 20 years old.
2. Diagnosed as patients suffered by skin tumor, brain tumor and breast tumor.

Exclusion Criteria:

1. Patients who can't speak and communicate with others.
2. Patients who can't make eventual and exact pathological assessment for his/her diseases.
3. Patients who only can fit for slicing tumor.
4. Removed tissues which obviously vary after severe ray radiation under microscopy observation.
5. Diameter of tumors are under 1 centimeter.
6. Breast carcinoma in situ.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anticpated the study population of tumor assessment:
  1. Skin cancer : 50.
  2. Brain tumor : 50.
  3. Breast cancer : 100.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The assessment between tumor cases and control cases | 5 years
  Do comparison with images acquired by our microscopy (with the whole-mount staining method) and bright field microscopy (with standard FFPE method) and do assessment to interpret tumor characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, National Taiwan University Hospital and College of Medicine, National Taiwan University, Taipei, Taiwan